CLINICAL TRIAL: NCT05026008
Title: A Randomized, Double-blind, Placebo-controlled, 2-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of SR1375 in Healthy Volunteers
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SR1375
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SR1375-101
Record Dates: First submitted 2021-08-18; First posted 2021-08-30 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SR1375 Capsule (Experimental): Ascending single and multiple doses of SR1375 capsules orally
  Interventions: Drug: SR1375
- Matching placebo (Experimental): Ascending single and multiple doses of placebo capsules orally
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: SR1375 — The subject will be orally administered by single and multiple doses of SR1375 capsules with 240 ml water
  Arms: SR1375 Capsule
Drug: Matching placebo — The subject will be orally administered by single and multiple doses of matching capsules with 240 ml water
  Arms: Matching placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2-part study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple ascending doses of SR1375 in healthy volunteers

DETAILED DESCRIPTION:
This study is a phase 1,randomized, double-blind, placebo-controlled, 2-part study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple ascending doses of SR1375 in healthy volunteers. The study is divided into two parts, Part A (single ascending dose [SAD]) and Part B (multiple ascending dose [MAD]). In Part A, the scheduled dose cohorts include 1, 3, 10, 30, 100, and 200 mg; in Part B, the planned dose range will be 5, 15, and 50 mg.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers will be included in the study if they satisfy all the following criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males (for both SAD and MAD stage) and female (only for MAD stage), 18 to 55 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2, with a body weight ≥ 50 kg at screening.
4. Use of tobacco or nicotine-containing products:
5. Medically healthy without clinically significant abnormalities at the screening visit, at check-in on Day -1 and pre-dose on Day 1.
6. Conventional 12-lead ECG recording in triplicate (the mean of triplicate measurements will be used to determine eligibility at the screening visit, on Day -1 and pre-dose on Day 1) consistent with normal cardiac conduction and function.
7. Have suitable venous access for blood sampling.
8. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

Volunteers will be excluded from the study if there is evidence of any of the following:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past three months determined by the Investigator to be clinically relevant.
2. Any history of malignant disease in the last 10 years (excluding completely treated cutaneous squamous cell or basal cell carcinoma).
3. Liver function test results (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gamma glutamyl transferase [GGT]) and bilirubin (total, conjugated and unconjugated) elevated more than 1.5-fold above the upper limit of normal (ULN).
4. Positive test results for active human immunodeficiency virus (HIV-1 and HIV-2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
5. Presence or having sequelae of gastrointestinal, liver (including Gilbert's syndrome), kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs. Exception: cholecystectomy is allowed.
6. History of substance abuse or alcohol abuse defined as >21 units of alcohol per week for males and >14 units of alcohol per week for females (for MAD cohorts only). One unit is equivalent to 8 g of alcohol: a half-pint (~285 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
7. Is an employee of an Investigator or Sponsor or an immediate relative of an Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
AE (Adverse Event) | Up to Day 32
  Incidence, type and severity and causality of AEs (including withdrawals due to safety or tolerability reasons)

SECONDARY OUTCOMES:
Plasma PK : Tmax | Up to Day 32
  Plasma PK : Time to Cmax (Tmax)
Plasma PK : Ctrough | Up to Day 32
  Plasma PK : Trough concentrations (Ctrough) (Part B only)
Plasma PK : AUC0-t | Up to Day 32
  Plasma PK : Area under the concentration-time curve from 0 to time of last quantifiable
Plasma PK : AUC0-∞ | Up to Day 32
  Plasma PK : Area under the concentration-time curve from t=0 to infinity (AUC0-∞)
Urine PK: Ae | Up to Day 4
  Urine PK: Cumulative amount of unchanged drug excreted in urine (Ae)
Urine PK: CLr | Up to Day 4
  Urine PK: Renal clearance (CLr)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Redfern, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No